CLINICAL TRIAL: NCT01031121
Title: Breath Carbon Monoxide and Cotinine as Biomarkers to Distinguish Smokers From Nonsmokers
Status: Completed | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909451; 09-DA-N451
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-10-22

CONDITIONS: Nicotine Dependence
Keywords: Cigarette Smoking; Biomarkers; Nicotine; Cotinine; Metabolites
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Background:

* Self-report and biochemical verification are used to determine smoking status in treatment trials and clinical research. Each method has merits and limitations that make it appropriate for particular situations. Participants who feel social pressure to report tobacco abstinence may provide unreliable self-reporting results. Biochemical verification using breath carbon monoxide (CO) is a more reliable indicator, but several biological and environmental factors (including exposure to secondhand smoke) can affect the sensitivity and specificity of breath CO measurement.
* An ideal biomarker of smoking status is cotinine, the major metabolite of nicotine. Cotinine levels found in blood, urine, and saliva can be used to distinguish between smokers and nonsmokers, as well as between light and heavy smokers. Researchers are interested in using cotinine assessments to develop suitable breath CO cutoff levels to categorize different types of smokers and nonsmokers for use in future research.

Objectives:

- To determine a breath carbon monoxide (CO) cutoff level that optimally discriminates between heavy and light smokers and nonsmokers who are and who are not exposed to environmental tobacco smoke.

Eligibility:

* Individuals between 18 and 64 years of age who fall into one of the following groups:
* current smokers reporting more than 10 cigarettes per day for at least 6 months
* current smokers reporting 10 or fewer cigarettes per day for at least 6 months
* nonsmokers reporting regular environmental exposure to tobacco smoke
* nonsmokers reporting limited or no exposure to tobacco smoke

Design:

* The study will involve a single outpatient session.
* Participants will provide breath CO, urine, and saliva samples, and will complete several smoking-related questionnaires on smoking history, current craving levels, and perceived level of nicotine dependence.

DETAILED DESCRIPTION:
Objective:

To determine a breath carbon monoxide (CO) cutoff level that optimally discriminates between heavy and light smokers and nonsmokers who are and who are not exposed to environmental tobacco smoke. Breath CO will be compared against cotinine concentration, which is the gold standard in verifying smoking status.

Study population:

The study will include four groups: 1) 60 smokers reporting > 10 cigarettes per day, 2) 60 smokers reporting less than or equal to 10 cigarettes per day, 3) 60 nonsmokers reporting regular environmental exposure to tobacco smoke, and 4) 60 nonsmokers reporting limited or no environmental exposure to tobacco smoke (total of 120 smokers and 120 nonsmokers).

Design:

Parallel groups design.

Outcome Measures:

1) breath CO; 2) semiquantitative salivary cotinine; 3) quantitative salivary nicotine, cotinine, and 3-hydroxycotinine; 4) semiquantitative urinary cotinine; 5) quantitative urinary nicotine, cotinine, norcotinine, and 3-hydroxycotinine; and 6) self-reported smoking variables.

ELIGIBILITY:
* INCLUSION CRITERIA:

For Smokers:

1. males and females 18-64 years old
2. smoking 1-10 cigarettes or > 10 cigarettes per day for the past 6 months

For Nonsmokers:

1. males and females 18-64 years old

EXCLUSION CRITERIA:

For Smokers:

1. current interest in reducing or quitting smoking
2. treatment for nicotine dependence in the past 3 months
3. use of nicotine replacement products, bupropion, or varenicline in the past 3 months
4. current use of tobacco products other than cigarettes
5. marijuana use greater than 5 times in past 14 days or use during 24 hours before session
6. chronic pulmonary disease
7. study investigator or subordinate staff

For Nonsmokers:

1. use of any tobacco or nicotine products in the past 3 months
2. marijuana use greater than 5 times in past 14 days or use during 24 hours before session
3. chronic pulmonary disease
4. study investigator or subordinate staff

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2009-06-08; Study Completion 2010-10-22

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Benowitz NL. Biomarkers of environmental tobacco smoke exposure. Environ Health Perspect. 1999 May;107 Suppl 2(Suppl 2):349-55. doi: 10.1289/ehp.99107s2349. PMID 10350520
- [Background] Bernert JT, Harmon TL, Sosnoff CS, McGuffey JE. Use of continine immunoassay test strips for preclassifying urine samples from smokers and nonsmokers prior to analysis by LC-MS-MS. J Anal Toxicol. 2005 Nov-Dec;29(8):814-8. doi: 10.1093/jat/29.8.814. PMID 16374940
- [Background] Chatkin J, Fritscher L, de Abreu C, Cavalet-Blanco D, Chatkin G, Wagner M, Fritscher C. Exhaled carbon monoxide as a marker for evaluating smoking abstinence in a Brazilian population sample. Prim Care Respir J. 2007 Feb;16(1):36-40. doi: 10.3132/pcrj.2007.00008. PMID 17297525